CLINICAL TRIAL: NCT01195571
Title: A Dose Escalation Study to Assess the Safety and Immunogenicity of Four Live Attenuated Human Cytomegalovirus(HCMV) Vaccines in Healthy Adults Without Prior Immunity.
Brief Title: Safety Study of Four Chimera Cytomegalovirus (CMV) Vaccines in Healthy Adult Males 30-50 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CMV Research Foundation (Other)
Collaborators: International AIDS Vaccine Initiative (Network)
Responsible Party: Principal Investigator, Stuart P. Adler, Principal Investigator, CMV Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Cytomegalovirus
MeSH Terms: interventions — mRNA-1647 cytomegalovirus vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccine administration (No Intervention): Each subject will receive on of four chimera CMV vaccines
  Interventions: Biological: cmv vaccine

INTERVENTIONS:
Biological: cmv vaccine — dose escalation study of 4 towne-toledo chimera vaccines
  Other Names: Towne vaccine; Toledo vaccine

SUMMARY:
The purpose of this research study is to test the safety and tolerability of four new investigational Cytomegalovirus (CMV) vaccines (Towne-Toledo 1, 2, 3, 4) in healthy male volunteers who are CMV negative. CMV is a common virus, infecting 50-80% of adults in the United States by the age of twenty-one. CMV does not usually cause illness in adults or children. However, CMV can be a cause of deafness and mental retardation in a child if a mother is infected during pregnancy. It also can be a serious illness in patients with impaired immunity (decreased ability to fight infection).

DETAILED DESCRIPTION:
A total of thirty six participants will be enrolled. The first 12 participants will be randomized into four groups. Four groups will receive one of the four investigational vaccines. The four investigational HCMV vaccine candidates will be administered subcutaneously to 3 volunteers at 10 pfu (the lowest dose to be used). The safety and tolerability of the four investigational HCMV vaccine candidates will be monitored closely for a period of 12 weeks following vaccination at this dose. Investigational vaccines that are found to be safe and well tolerated at a dose of 10pfu will be administered to 3 additional individuals at 102 pfu and then at 103 pfu. Safety and tolerability will be evaluated at each dose level by monitoring clinical signs and symptoms, laboratory parameters and virus detection in the blood, urine, and saliva. After the 12-week safety-monitoring period, participants will be followed for the remainder of one year to assess long-term safety and immunogenicity of the investigational vaccines.

ELIGIBILITY:
Inclusion Criteria:

* a) Healthy male adult, between the ages of 30 to 50 years with no children <18 years of age at home and in a stable sexual or household relationship with an individual who must be CMV seropositive, non-pregnant, not planning a pregnancy within one year and not currently breastfeeding.

  b) HCMV seronegative. c) HIV seronegative. d) Hepatitis B surface antigen negative. e) No evidence of active hepatitis C infection by serologic evaluation. f) HCMV culture negative (to be determined by shell vial or routine culture of urine, blood and saliva collected at the screening visit).

  g) Agrees to abstain from sex or to use condoms during intercourse for 52 weeks following vaccination.

  h) Available by telephone or pager for one year following vaccination. i) Willing and able to comply with the requirements of the protocol and to properly complete participant diaries.

  j) Signed informed consent and completed social/demographic questionnaire. k) Willing to forego blood, bone marrow or whole organ donation for 1year post vaccination.

  l) Willing to forego enrollment in studies of other investigational agents for one year following vaccination.

Exclusion Criteria:

1. History of immunodeficiency or any ongoing serious disease such as cancer, autoimmune disease, HIV infection, chronic renal failure (whether or not on dialysis), or diabetes.
2. Significant acute or chronic infection at the time of vaccination.
3. Household contact with an immunosuppressed individual.
4. History of anaphylaxis or severe vaccine reaction.
5. Vaccination with a live vaccine within the past month or an inactivated vaccine within two weeks prior to vaccination, or plan to receive any vaccine within two months following vaccination.
6. Seropositive sexual partner who desires to become pregnant within one year following vaccination, currently is pregnant, or is currently breast feeding.
7. Has a close contact who is CMV seronegative or who is ineligible or chooses not to participate in the study.
8. Received blood products in proceeding three months or expects to receive blood products within the following year.
9. A childcare provider.
10. A health care provider who routinely comes in contact with pregnant women or immunologically compromised persons.
11. Any condition which, in the opinion of the investigator, may interfere with adherence to the protocol or make it inadvisable to enroll the participant.
12. Currently participating in a study of any other experimental or investigational agent, or has participated in such a study within a month of vaccination.
13. Previous vaccination with an investigational HCMV vaccine.
14. Treatment with excluded antiviral or immunosuppressive drugs (Appendix D) within one month prior to vaccination.
15. Expected use of antiviral or immunosuppressive agents within two months following vaccination.
16. Any screening safety laboratory value that is outside normal limits of the laboratory normal range (screening laboratory tests may be repeated if minor abnormalities or possible laboratory errors are noted).

    -

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety | 2 years
  To evaluate the safety and tolerability, in adults without prior HCMV immunity (seronegative), of four live attenuated HCMV investigational vaccines at each of three dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart P Adler, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Adler SP, Manganello AM, Lee R, McVoy MA, Nixon DE, Plotkin S, Mocarski E, Cox JH, Fast PE, Nesterenko PA, Murray SE, Hill AB, Kemble G. A Phase 1 Study of 4 Live, Recombinant Human Cytomegalovirus Towne/Toledo Chimera Vaccines in Cytomegalovirus-Seronegative Men. J Infect Dis. 2016 Nov 1;214(9):1341-1348. doi: 10.1093/infdis/jiw365. Epub 2016 Aug 11. PMID 27521362